CLINICAL TRIAL: NCT03370393
Title: Prevention of Adolescent Risky Behaviors: Neural Markers of Intervention Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Uma Rao, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20173439; R01DA040966 (NIH)
Record Dates: First submitted 2017-12-01; First posted 2017-12-12 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Risk-Taking; Adolescent Behavior
Keywords: Reward-drive; Cognitive-control
MeSH Terms: conditions — Risk-Taking; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: The families will be randomized to Pathways for African Americans' Success (PAAS) intervention program or a wait-list condition (1:1 ratio) for 6 weeks. The wait-list group has the option to participate in the PAAS program at the end of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pathways for African-Americans' Success (Experimental): Subjects will complete a 6-week Pathways for African-Americans' Success (PAAS) intervention. This is a weekly, 1.5 hour/session, family intervention for 6 weeks.
  Interventions: Behavioral: Pathways for African-Americans' Success (PAAS)
- Wait-list (No Intervention): Subjects will be on waiting list for active intervention and will receive the PAAS intervention at the end of the study (same as active intervention).

INTERVENTIONS:
Behavioral: Pathways for African-Americans' Success (PAAS) — PAAS is a 6-week, technology-delivered, family-based youth risk intervention program. PAAS includes 6 sessions for parents and youth, and joint sessions in which they both engage on the same computer to integrate and practice the skills they have just learned in their separate sessions. Each session includes a review, a virtual discussion, and observing and interacting with four parent and four youth Avatars that reflect phenotypes of African Americans (AA), with voice-overs by AA parents and youth. Videos portraying family interactions and intrapersonal processes are integrated into each session to convey key points of the intervention along with interactive activities to promote skill-building and to reinforce learning. PAAS also includes a technology tutorial and an introductory session.
  Arms: Pathways for African-Americans' Success

SUMMARY:
Adolescence is a time of biological and behavioral changes that can lead to risky and dangerous behaviors, and African-American youth are highly vulnerable to the consequences of risky behavior, including HIV/AIDS and violence, leading to premature death. The investigators previously showed that an intervention program reduces HIV-risk vulnerability behaviors in many African-American youth. The investigators aim to measure how the program affects different regions of the brain in order to better prevent or reduce such risky behaviors among African-American youth.

DETAILED DESCRIPTION:
Adolescence is a time of dramatic biological, behavioral and social changes. It is one of the healthiest periods of the life-span, yet morbidity and mortality rates increase 200%, often attributed to natural tendencies to explore and take risks that increase vulnerability to risky and dangerous behaviors. Rapid advances in developmental neuroscience are revealing new insights into how biology and social context interact to increase adolescents' risk-taking behavior which is attributed to a temporal disassociation between maturational changes in two distinct neural systems: "socio-emotional" (reward) and "cognitive-control" (self-regulation). The socio-emotional system is stimulated by a rapid increase in dopaminergic activity at puberty, which influences reward-seeking behavior. This increase in reward-seeking precedes the maturation of the cognitive-control system and its connections to the reward system. This proposal aims to apply these new insights on neurobiology of adolescents' responses to alcohol/drug use and sex-related risk opportunities by examining brain changes in response to a theoretically-based and empirically-tested prevention program that targets risky behavior in African-American youth during pubertal transition. This racial group is disproportionately affected by the high morbidity and mortality associated with HIV-related risky behaviors and exemplifies a significant health disparity in our society. The intervention was designed on the basis of developmental issues and socio-cultural contextual processes germane to African-American families, and has been shown in randomized controlled trials to delay/deter HIV-related risky behaviors in this vulnerable population. This proposal extends the efficacy studies of the intervention by using functional magnetic resonance imaging to quantify the biological changes in response to the intervention. Identifying neural substrates of the intervention can facilitate refinement of the program by focusing on the components that are most effective in changing behavioral and neural circuitry and also aid in the development of new interventions for subgroups of youth that don't have a positive outcome. Using a randomized controlled design, the investigators will assess the neural substrates of risk-taking and risk-avoidant behavior before and after the 6-week computer-interactive, family-based intervention in 11-13 year-old African-American youth. Psychological processes shown to mediate the intervention effects on behaviors that dissuade alcohol and drug use and sexual onset (i.e. reward-drive and cognitive-emotional self-regulation) will be assessed at baseline and 3 months post-intervention. Based on prior studies that reported observable brain changes in response to psychosocial interventions, the investigators' hypothesis is that a positive response to the intervention will be associated with greater functional connectivity changes between the socio-emotional (reward-drive) and cognitive-control (self-regulation) components of the neural circuitry compared to the control condition, both at rest and during task-performance. They also postulate that these neural changes will mediate the intervention's positive effects on psychological processes involved in youth's decision to avoid HIV-risk vulnerability behaviors in the service of long-term personal goals and positive health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subject is of African-American racial status (self-reported)
* Subject can speak and read English
* Subject and parent/legal guardian agree to participate in the 6-week PAAS program
* Subject and parent/legal guardian agree to complete all assessments
* Subject must meet MRI safety eligibility

Exclusion Criteria:

* Subject has a major medical problem (e.g. neurological disorders)
* Subject is on medication(s) that affects the central nervous system
* Subject has behavioral/emotional problems at a clinical level (parent and/or youth report)
* Subject is pregnant or suspected of being pregnant (based on pregnancy test)
* Subject is color-blind
* Subject has claustrophobia
* Subject has metallic implants
* Subject drinks alcohol in the week prior to entry into the study (based on urine drug screen)
* Subject uses drugs in the week prior to entry into the study (based on urine drug screen)

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uma Rao, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pathways for African-Americans' Success: Subjects completed a 6-week Pathways for African-Americans' Success (PAAS) intervention. This is a weekly, 1.5 hour/session, family intervention for 6 weeks.
  Pathways for African-Americans' Success (PAAS): PAAS is a 6-week, technology-delivered, family-based youth risk intervention program. PAAS includes 6 sessions for parents and youth, and joint sessions in which they both engage on the same computer to integrate and practice the skills they have just learned in their separate sessions. Each session includes a review, a virtual discussion, and observing and interacting with four parent and four youth Avatars that reflect phenotypes of African Americans (AA), with voice-overs by AA parents and youth. Videos portraying family interactions and intrapersonal processes are integrated into each session to convey key points of the intervention along with interactive activities to promote skill-building and to reinforce learning. PAAS also includes a technology tutorial and an introductory session.
- Wait-list: Subjects were on a wait list for active intervention and received the PAAS intervention at the end of the study (same as active intervention).
Period: Overall Study
Arm/Group | Pathways for African-Americans' Success | Wait-list
Started | 86 | 60
Completed | 71 | 50
Not Completed | 15 | 10
Not completed — Lost to Follow-up | 15 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pathways for African-Americans' Success | Wait-list | Total
Number analyzed (Participants) | 86 | 60 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 86 | 60 | 146
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.56 (1.0) | 12.57 (1.0) | 12.56 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 26 | 64
  Male | 48 | 34 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 86 | 60 | 146
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Southern California (participants were recruited across Southern California, including Los Angeles, Orange, San Bernadino and San Diego counties)
  Participants
    United States | 86 | 60 | 146
Emotion regulation [Mean (Standard Deviation); unit: T score] — Emotional regulation was assessed through parent and youth self-reported questionnaires using the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2). T scores, normed for age and sex are available. T-score standardizes an individual's executive functioning difficulties relative to peers. For example, 50 is the population mean and a standard deviation of 10. Higher scores indicate more significant problems. Scores below 60 are within normal limits; 60-64: subclinical difficulties; 65-69: mildly elevated; 70-74: moderately elevated; and 75 or above: highly elevated
  T score | 54.43 (12.23) | 52.02 (10.15) | 53.44 (11.45)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Emotional Regulation
Description: Emotional regulation was assessed through parent and youth self-reported questionnaires using the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2). T scores, normed for age and sex are available. T-score standardizes an individual's executive functioning difficulties relative to peers. For example, 50 is the population mean and a standard deviation of 10. Higher scores indicate more significant problems. Scores below 60 are within normal limits; 60-64: subclinical difficulties; 65-69: mildly elevated; 70-74: moderately elevated; and 75 or above: considered highly elevated, suggesting significant difficulties in emotion regulation. These questionnaires were administered at baseline (before intervention) and 3 months post-intervention. Because parent report may be less biased regarding youth's regulation, we used parent data for analysis. Data imputation was done for missing data.
Time Frame: 18 weeks (from pre-intervention to 3-months after post-intervention)
Measure: Mean (Standard Deviation); unit: T Score
Groups:
- Wait-list: Subjects were on waitlist for active intervention and were offered the PAAS intervention at the end of the study (same as active intervention).
Arm/Group | Pathways for African-Americans' Success | Wait-list
Number analyzed (Participants) | 86 | 60
T Score
  Pre-intervention (baseline) | 54.43 (12.23) | 52.02 (10.15)
  Post-intervention (3-month follow-up after 6-week intervention) | 54.47 (13.74) | 60.77 (16.76)
Statistical Analysis 1: Comparison: Pathways for African-Americans' Success vs Wait-list; Test type: Equivalence — Two-way repeated measures analysis. If the group*time interaction is positive, then the groups differ with respect to intervention effects; p = 0.003, Wilk's Lambda; Mean Difference (Final Values) = 9.40

2. Secondary Outcome: Changes in Cognitive Regulation
Description: Cognitive regulation was assessed through parent and youth self-reported questionnaires using the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2). T scores, normed for age and sex are available. T-score standardizes an individual's executive functioning difficulties relative to peers. For example, 50 is the population mean and a standard deviation of 10. Higher scores indicate more significant problems. Scores below 60 are within normal limits; 60-64: subclinical difficulties; 65-69: mildly elevated; 70-74: moderately elevated; and 75 or above: considered highly elevated, suggesting significant difficulties in cognitive regulation. These questionnaires were administered at baseline (before intervention) and 3 months post-intervention. Because parent report may be less biased regarding youth's regulation, we used parent data for analysis. Data imputation was done for missing data.
Time Frame: 18 weeks (from pre-intervention to 3-months after post-intervention)
Population: One participant did not complete this section
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Pathways for African-Americans' Success | Wait-list
Number analyzed (Participants) | 86 | 59
T Score
  Pre-intervention (baseline) | 55.41 (10.71) | 54.51 (10.52)
  post-intervention (3-month follow-up after intervention) | 51.81 (20.94) | 55.66 (18.44)
Statistical Analysis 1: Comparison: Pathways for African-Americans' Success vs Wait-list; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.45, Wilk's Lambda; Mean Difference (Final Values) = 0.566

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline (pre-treatment) visit until 3 months post-intervention visits
Description: Serious and non-serious adverse events
Arm/Group | Pathways for African-Americans' Success | Wait-list
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/60
Other Adverse Events (participants affected / at risk) | 0/86 | 0/60

LIMITATIONS AND CAVEATS:
Trial was completed successfully.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT03370393/Prot_SAP_004.pdf
  • Informed Consent Form (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT03370393/ICF_003.pdf